CLINICAL TRIAL: NCT01028027
Title: A Clinical Safety and Efficacy Evaluation of Zylet® Versus Tobradex in the Treatment of Blepharokeratoconjunctivitis
Brief Title: Loteprednol and Tobramycin Versus Tobramycin and Dexamethasone, in the Treatment of Blepharokeratoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 617
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2011-09-15 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Conjunctivitis; Keratitis; Blepharitis
Keywords: Blepharokeratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis; Keratitis; Blepharitis | interventions — Loteprednol Etabonate; Tobramycin; Dexamethasone; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol and tobramycin (Experimental): Loteprednol etabonate and tobramycin ophthalmic suspension
  Interventions: Drug: Loteprednol and tobramycin
- Tobramycin and dexamethasone (Active Comparator): Tobramycin and dexamethasone ophthalmic suspension
  Interventions: Drug: Tobramycin and dexamethasone

INTERVENTIONS:
Drug: Loteprednol and tobramycin — Loteprednol etabonate and tobramycin ophthalmic suspension administered to study eye 4 times a day (QID) for 14 days.
  Other Names: Zylet
  Arms: Loteprednol and tobramycin
Drug: Tobramycin and dexamethasone — Tobramycin and dexamethasone ophthalmic suspension administered to study eye 4 times a day (QID) for 14 days.
  Other Names: Tobradex
  Arms: Tobramycin and dexamethasone

SUMMARY:
This study is to evaluate the safety and efficacy of loteprednol etabonate [LE] and tobramycin ophthalmic suspension versus tobramycin and dexamethasone ophthalmic suspension in the treatment of ocular inflammation associated with blepharokeratoconjunctivitis (BKC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of BKC in at least one eye
* Subjects must be willing to discontinue contact lens use for the duration of the study
* Subjects who are able and willing to comply with all treatment and follow- up/study procedures.

Exclusion Criteria:

* Subjects participating in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.
* Subjects who have any uncontrolled systemic disease or debilitating disease.
* Subjects who have a known hypersensitivity to the study drugs or their components (including benzalkonium chloride) or contraindications to tobramycin or ocular corticosteroids.
* Subjects who use any topical or systemic ophthalmic medications listed as disallowed in the study protocol, within the specified time frame prior to Visit 1.
* Subjects who have a disease or conditions which the Investigator determines could interfere with the safety and efficacy evaluations of the study drug.
* Subjects having ocular surgery (including laser surgery) in either eye within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Chu, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Inc, Singapore, Singapore

REFERENCES:
- [Derived] Chen M, Gong L, Sun X, Gu Y, He X, Qu J, Wang L, Zhang M, Zhong X. A multicenter, randomized, parallel-group, clinical trial comparing the safety and efficacy of loteprednol etabonate 0.5%/tobramycin 0.3% with dexamethasone 0.1%/tobramycin 0.3% in the treatment of Chinese patients with blepharokeratoconjunctivitis. Curr Med Res Opin. 2012 Mar;28(3):385-94. doi: 10.1185/03007995.2012.659723. Epub 2012 Feb 7. PMID 22256909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at seven sites, by seven Investigators in the People's Republic of China. First participant was enrolled 10/21/2009 and last participant visit was 2/9/2010.
Pre-assignment Details: A total of 357 participants with clinically diagnosed blepharokeratoconjunctivitis (BKC) in at least one eye were enrolled. 328 participants completed the study.
Groups:
- Loteprednol and Tobramycin: Loteprednol etabonate 0.5% and tobramycin 0.3% ophthalmic suspension. Participants will instill one or two drops of study drug topically in the affected eye(s), at approximately four hour intervals, QID, for 14 days.
- Tobramycin and Dexamethasone: Tobramycin 0.3% and dexamethasone 0.1% ophthalmic suspension. Participants will instill one or two drops of study drug topically in the affected eye(s), at approximately four hour intervals, QID, for 14 days.
Period: Overall Study
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Started | 180 | 177
Completed | 164 | 164
Not Completed | 16 | 13
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 4 | 7
Not completed — Protocol Violation | 3 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone | Total
Number analyzed (Participants) | 180 | 177 | 357
Age Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (13.63) | 41.72 (13.54) | 41.26 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 113 | 236
  Male | 57 | 64 | 121
Region of Enrollment [Number; unit: participants]
  Singapore | 180 | 177 | 357

OUTCOME MEASURES:

1. Primary Outcome: Signs and Symptoms Composite Score - Change From Baseline to Day 15 - PP Population
Description: The change from baseline (CFB) to Day 15 (Visit 4) in the ocular signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score. Per protocol population (PP).
Time Frame: Baseline, Day 15
Population: The PP population was the population used for the primary efficacy analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Number analyzed (Participants) | 156 | 152
Scores on a scale | -11.63 (4.56) | -12.41 (4.71)

2. Secondary Outcome: Signs and Symptoms Composite Score - Change From Baseline to Day 15 - ITT Population
Description: The CFB to Day 15 in the signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score. ITT population
Time Frame: Baseline, Day 15
Population: The ITT population was used in this secondary efficacy parameter.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Number analyzed (Participants) | 164 | 165
Score on a scale | -11.64 (4.55) | -11.98 (4.95)

3. Secondary Outcome: Signs and Symptoms Composite Score - Change From Baseline to Day 8 - PP Population
Description: The CFB to Day 8 (Visit 3) in the signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score.
Time Frame: Baseline, Day 8
Population: The PP population was used for this secondary efficacy parameters.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Number analyzed (Participants) | 155 | 150
Score on a scale | -9.20 (3.94) | -10.21 (4.23)

4. Secondary Outcome: Signs and Symptoms Composite Score - Change From Baseline to Day 8 - ITT Population
Description: The CFB to Day 8 in the signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score. ITT population
Time Frame: Baseline, Day 8
Population: The ITT population was used in this secondary efficacy parameter.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Number analyzed (Participants) | 172 | 171
Score on a scale | -8.91 (4.24) | -9.96 (4.27)

5. Secondary Outcome: Signs and Symptoms Composite Score Change From Baseline to Day 3 - PP Population
Description: The CFB to Day 3 in the signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score. PP population.
Time Frame: Baseline, Day 3
Population: The PP population was used for this secondary efficacy parameters.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Number analyzed (Participants) | 155 | 152
Score on a scale | -5.66 (3.46) | -5.98 (3.68)

6. Secondary Outcome: Signs and Symptoms Composite Score Change From Baseline to Day 3 - ITT Population
Description: The CFB to Day 3 in the signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score. ITT population.
Time Frame: Baseline, Day 3
Population: The ITT population was used for this secondary efficacy parameters.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Number analyzed (Participants) | 177 | 176
Score on a scale | -5.54 (3.48) | -5.92 (3.69)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Loteprednol and Tobramycin | Tobramycin and Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/177
Other Adverse Events (participants affected / at risk) | 16/177 | 36/177
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol and Tobramycin (N=177) | Tobramycin and Dexamethasone (N=177)
Increased IOP (Eye disorders) | 16 (52) | 36 (52) — Overall IOP change from baseline >5mmHg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.